CLINICAL TRIAL: NCT03998800
Title: The Effect of L-arginine and L-citrulline Supplementation on Endurance Performance and Mitochondrial Respiration
Brief Title: Effects of L-arginine and L-citrulline Supplementation on Muscle Respiration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Collaborators: Kyowa Hakko Bio Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Stephen Bailey, Lecturer in Sport ad Exercise Nutrition, Loughborough University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: R19-P010
Record Dates: First submitted 2019-06-18; First posted 2019-06-26 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Dietary Exposure
Keywords: Endurance performance; Mitochondrial function; L-arginine; L-citrulline; Healthy males
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Intervention Model Description: Allocation: Randomized Endpoint Classification: Efficacy Study Intervention Model: Crossover Assignment Masking: Double Blind (Subject, Investigator)
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- L-arginine and L-citrulline (Experimental): 10 days of supplementation with 1.5 g of L-arginine and 1.5 g of L-citrulline per day
  Interventions: Dietary Supplement: Dietary Supplement; Behavioral: Endurance exercise on a cycle ergometer
- L-arginine (Experimental): 10 days of supplementation with 3 g of L-arginine per day
  Interventions: Dietary Supplement: Dietary Supplement; Behavioral: Endurance exercise on a cycle ergometer
- Placebo (corn-starch) (Placebo Comparator): 10 days of supplementation with corn-starch
  Interventions: Dietary Supplement: Dietary Supplement; Behavioral: Endurance exercise on a cycle ergometer

INTERVENTIONS:
Dietary Supplement: Dietary Supplement — Dietary Supplement: L-arginine and L-citrulline supplement, L-arginine supplement, or placebo supplement (corn-starch) Subjects will complete 3 individual 10 day supplementation periods, separated by washout periods of approximately 2 weeks.
Behavioral: Endurance exercise on a cycle ergometer — On day 10 of each supplementation period, subjects will complete a performance test on a cycle ergometer to investigate their endurance performance.

SUMMARY:
The objective of this trial is to determine the effects of dietary supplementation with the amino acids, L-arginine and L-citrulline, on endurance performance and mitochondrial respiration in healthy men compared to supplementation with L-arginine alone and a placebo supplement.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, cross over trial of L-arginine and L-citrulline supplementation, L-arginine supplementation alone and placebo supplementation in healthy men. The intervention period will be 8-11 weeks for each participant and a minimum of 15 individuals will be recruited and enrolled to complete the trial. Subjects will complete the experimental protocol described below over 3 individual 10 day supplementation periods, separated by washout periods of approximately 2 weeks. Subjects will ingest corn-starch as a placebo, L-arginine (3g/day) or L-arginine (1.5 g/day) + L-citrulline (1.5g/day). On day 7 of the supplementation period, a skeletal muscle biopsy and blood sample will be obtained from the subjects to investigate mitochondrial function and blood amino acid and nitric oxide levels. On day 10 of the supplementation period, subjects will complete a performance test on a cycle ergometer to investigate their endurance performance. These assessments will be performed to determine the effects of co-ingesting L-arginine and L-citrulline compared to L-arginine alone and placebo administration.

ELIGIBILITY:
Inclusion Criteria:

* healthy male, 18-40 years of age
* recreationally-active
* healthy BMI (≥18.5 and ≤24.9 kg/m2)

Exclusion Criteria:

* participating in other studies currently or in the past two months or has an intention to participate in other studies over the period of this study
* history of gastric, digestive, cardiovascular, renal disease or any other orthopaedic diseases related to motor organs
* lidocaine allergy
* use of medication that may affect study measures
* contraindication to the biopsy procedures
* on medications that affect the immune system
* on Aspirin or other drugs known to prolong bleeding
* smoker
* user of dietary supplements currently or in the past one month
* a heavy drinker

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Change in Endurance performance on a cycle ergometer between L-arginine supplementation and placebo supplementation | 8-11 weeks
  On day 10 of the supplementation periods, subjects will complete a performance test on a cycle ergometer to investigate their endurance performance
Change in Endurance performance on a cycle ergometer between L-arginine + L-citrulline supplementation and placebo supplementation | 8-11 weeks
  On day 10 of the supplementation periods, subjects will complete a performance test on a cycle ergometer to investigate their endurance performance
Changes of mitochondrial function in skeletal muscle between L-arginine supplementation and placebo supplementation | 8-11 weeks
  On day 7 of the supplementation periods, a skeletal muscle biopsy sample will be obtained from subjects to investigate mitochondrial function.
Changes of mitochondrial function in skeletal muscle between L-arginine + L-citrulline supplementation and placebo supplementation | 8-11 weeks
  On day 7 of the supplementation periods, a skeletal muscle biopsy sample will be obtained from subjects to investigate mitochondrial function.

SECONDARY OUTCOMES:
Changes of amino acid and nitric oxide biomarkers levels in plasma between L-arginine supplementation and placebo supplementation | 8-11 weeks
  On days 7 and 10 of the supplementation periods, a venous blood sample will be obtained from subjects to investigate amino acid and nitric oxide biomarkers levels in plasma.
Changes of amino acid and nitric oxide biomarkers levels in plasma between L-arginine + L-citrulline supplementation and placebo supplementation | 8-11 weeks
  On days 7 and 10 of the supplementation periods, a venous blood sample will be obtained from subjects to investigate amino acid and nitric oxide biomarkers levels in plasma.
Changes in muscle oxygenation between L-arginine supplementation and placebo supplementation | 8-11 weeks
  On day 10 of the supplementation periods, skeletal muscle oxygenation will be assessed using near-infrared spectroscopy to reveal the tissue saturation index during exercise.
Changes in muscle oxygenation between L-arginine + L-citrulline supplementation and placebo supplementation | 8-11 weeks
  On day 10 of the supplementation periods, skeletal muscle oxygenation will be assessed using near-infrared spectroscopy to reveal the tissue saturation index during exercise.
Changes in subjective feeling during and after exercise between L-arginine supplementation and placebo supplementation | 8-11 weeks
  On day 10 of the supplementation period, subjective feeling during (using the 6-20 ratings of perceived exertion scale) and after (using a 100 mm visual analogue scale where 0 mm = no pain and 100 m = maximal pain) exercise will be assessed. Subjective feeling will also be assessed on the morning of day 11 of each supplementation period.
Changes in subjective feeling during and after exercise between L-arginine + L-citrulline supplementation and placebo supplementation | 8-11 weeks
  On day 10 of the supplementation period, subjective feeling during (using the 6-20 ratings of perceived exertion scale) and after (using a 100 mm visual analogue scale where 0 mm = no pain and 100 m = maximal pain) exercise will be assessed. Subjective feeling will also be assessed on the morning of day 11 of each supplementation period.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Bailey, PhD, Principal Investigator — Lecturer
Locations (1):
- School of Sport, Exercise and Health Sciences, Loughborough, Leicester, United Kingdom